CLINICAL TRIAL: NCT02689453
Title: A Phase I Study of Subcutaneous Recombinant Human IL-15 (S.C. Rhil-15) and Alemtuzumab for Patients With Refractory or Relapsed Chronic and Acute Adult T-Cell Leukemia (ATL)
Brief Title: Subcutaneous Recombinant Human IL-15 (s.c. rhIL-15) and Alemtuzumab for People With Refractory or Relapsed Chronic and Acute Adult T-cell Leukemia (ATL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160062; 16-C-0062
Record Dates: First submitted 2016-02-20; First posted 2016-02-24 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: T-Cell Lymphoma Relapsed; Adult T-Cell Leukemia (ATL); Peripheral T-Cell Lymphoma (PTCL); Cutaneous T Cell Lymphoma (CTCL); T-Cell Prolymphocytic Leukemia
Keywords: T-cell Lymphoproliferative Disorder; CD4/CD25 Expressing T-cells in Blood and Lymphoid Tissues; Anti-CD52 Monoclonal Antibody; Antibody Dependent Cellular Cytotoxicity
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Leukemia, Prolymphocytic, T-Cell | interventions — Interleukin-15; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1A-Interleukin 15 (IL-15) Followed by Alemtuzumab (Experimental): IL-15 for 10 doses over two weeks followed by alemtuzumab for 4 weeks per dosing schema to determine the maximum tolerated dose (MTD)
  Interventions: Biological: IL-15 plus; Biological: alemtuzumab
- 1B - Interleukin-15 (IL-15) Followed by Alemtuzumab at the Maximum Tolerated Dose (Experimental): IL-15 for 10 doses over two weeks followed by alemtuzumab for 4 weeks at the maximum tolerated dose (MTD)
  Interventions: Biological: IL-15 plus; Biological: alemtuzumab

INTERVENTIONS:
Biological: IL-15 plus — Recombinant Human IL-15 (subcutaneous (s.c.) rhIL-15) by s.c. injection Monday-Friday over two weeks.
  Other Names: Interleukin-15
Biological: alemtuzumab — Alemtuzumab three times a week for a total of 4 weeks of alemtuzumab treatment.
  Other Names: Campath

SUMMARY:
Background:

Adult T-cell leukemia (ATL) is a rare blood cancer. Researchers want to see if a combination of two drugs - recombinant human interleukin 15 (rhIL-15) and alemtuzumab - is a better treatment for ATL.

Objectives:

To test if giving rhIL-15 combined with alemtuzumab improves the outcome of therapy for ATL. Also, to determine the safe dose of this combination and identify side effects and effects on the immune system.

Eligibility:

Adults 18 years and older with chronic or acute ATL who have not been helped by other treatments.

Design:

Participants will be screened with tests that are mostly part of their usual cancer care. They will sign a separate consent form for this.

Weeks 1 and 2: Participants will have a total of 10 visits. They will:

* Get rhIL-15 under the skin by needle.
* Have a physical exam and vital signs measured.
* Give blood samples.
* Answer questions about their health and their medicines.

Week 3: Participants will stay in the clinic. They will:

* Get alemtuzumab infusions in a vein through a small catheter on days 1, 2, 3, and 5.
* Take medicines to decrease side effects.
* Have a computed tomography (CT) scan to evaluate the treatment.
* Have a physical exam and vital signs measured.
* Give blood samples.

Answer questions about their health and medicines.

Weeks 4, 5, and 6 will repeat week 3, without the CT scan. Some patients will just have outpatient visits these weeks.

After treatment, participants will have follow-up visits every few months for up to 2 years. At these visits, participants will give blood samples and have CT scans.

DETAILED DESCRIPTION:
Background:

* A previous trial alemtuzumab (CAMPATH-1) in patients with chronic, acute and lymphomatous subtype HTLV-1 associated ATL showed appreciable initial activity but no clear long-term impact.
* Antibody dependent cellular cytotoxicity (ADCC) with polymorphonuclear neutrophils (PMNs), monocytes and natural killer (NK) cells acting as the effector cells is alemtuzumab s primary in vivo mechanism of action for depleting malignant leukemic or lymphomatous cells.
* The immunologic effects of Interleukin-15 (IL-15), a stimulatory cytokine that promotes the differentiation and activation of NK cells, monocytes and long-term cluster of differentiation 8 (CD8+) memory Tcells, has been assessed in several phase I trials in cancer patients.
* Administration of recombinant human (rh) IL-15 as an intravenous bolus (IVB), continuous intravenous infusion (CIV) or subcutaneous injections (SC) into adult cancer patients has produced 5 to 50 fold expansion in the number of circulating NK cells at well tolerated doses in these patients.
* Preclinical murine lymphoid malignancy models have shown efficacy from the administration of IL-15 and monoclonal antibodies, with improved survival compared to controls.

Objective:

-To determine the safety, toxicity profile and the maximum tolerated dose (MTD) of s.c. rhIL-15 in combination with standard three times per week IV alemtuzumab treatment.

Eligibility:

* Age greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 1
* Diagnosis of adult T-cell leukemia (Human T-cell lymphotropic virus type 1 (HTLV-1) associated, chronic or acute), peripheral T-cell lymphoma (angioimmunoblastic, hepatosplenic, or not otherwise specified), cutaneous T-cell lymphoma (Stage III or IV, with leukemia involvement or erythrodemia), or T-cell prolymphocytic leukemia (T-PLL)
* Measurable or evaluable disease
* Adequate organ and bone marrow function as defined in the protocol.

Design:

* This is a single institution nonrandomized Phase I dose escalation study evaluating increasing doses of subcutaneous (SC) rhIL-15 in combination with alemtuzumab using a standard 3 + 3 dose escalation.
* Treatment will include s.c. rhIL015 daily Monday-Friday (M-F) weeks 1 and 2 (dose levels 0.5- 2 mcg/kg/dose), followed by intravenous (IV) alemtuzumab beginning in week 3 (escalating doses followed by standard dosing in weeks 4-6).
* Up to 30 patients will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria

* Age greater than or equal to 18 years; no upper age limit.
* Patients diagnosed with a leukemia or lymphoma as follows:

  * Chronic or acute leukemia forms of Human T-cell lymphotropic virus type 1 (HTLV-1) associated adult T-cell leukemia;
  * Peripheral T-cell lymphoma (angioimmunoblastic, hepatosplenic, or not otherwise specified); or,
  * Cutaneous T-cell lymphoma stage III or IV with circulating monoclonal cells (B1 or B2) and/or erythrodermia (T4)
  * T-cell prolymphocytic leukemia (T-PLL)

NOTE: Diagnosis must be validated by the Pathology Department, National Cancer Institute (NCI).

-Patients must have measurable or evaluable disease.

NOTE: All patients with greater than 10% abnormal cluster of differentiation 4 (CD4+) homogeneous cluster of differentiation 3 (CD3) low strongly cluster of differentiation 25 (CD25+) expressing cells, or greater than 5% Szary cells/T-PLL, among the peripheral blood mononuclear cells (PBMCs) in the peripheral blood will be deemed to have evaluable disease.

* Abnormal T cells must be cluster of differentiation 52 (CD52+) as assessed by flow cytometry or immunohistochemistry.
* Patients must have a life expectancy of greater than or equal to 2 months.
* Patients must have been refractory or relapsed following front line therapy for Adult T-cell Leukemia (ATL); those with cutaneous T-cell lymphoma (CTCL) or peripheral T-cell lymphoma (PTCL) who have cluster of differentiation 30 (CD30+) disease must have progressed during or after treatment with brentuximab vedotin, or are unable to receive treatment due to allergy or intolerance.
* Patients must have recovered to less than grade 1 or to baseline from toxicity of prior chemotherapy or biologic therapy and must not have had major surgery, chemotherapy, radiation or biologic therapy within 2 weeks prior to beginning treatment. NOTE: Exceptions to this include events not considered to place the subject at unacceptable risk of participation in the opinion of the PI (e.g., alopecia).
* Carbon monoxide diffusing capacity alveolar volume (DLCO/VA) and forced expiratory volume (FEV) 1.0 > 50% of predicted on pulmonary function tests.
* Adequate laboratory parameters, as follows:

  * Serum creatinine of less than or equal to 1.5 x the upper limit of normal
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x the upper limit of normal
* Absolute neutrophil count greater than or equal to 1,500/mm^3 and platelets greater than or equal to 100,000/mm^3.
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 1.
* Patients must be able to understand and sign an Informed Consent Form.
* All patients must use adequate contraception during participation in this trial and for 4 months following completing therapy.

EXCLUSION CRITERIA:

* Patients who have received any systemic corticosteroid therapy within 4 weeks prior to the start of therapy, or 12 weeks if given to treat graft versus host disease (GVHD), with the exception of physiological replacement doses of cortisone acetate or equivalent.
* Patients who have undergone allogeneic stem cell transplantation and have required systemic treatment for GVHD (including but not limited to oral or parenteral corticosteroids, ibrutinib, and extracorporeal phototherapy) within the last 12 weeks
* Clinical evidence of (parenchymal or meningeal) central nervous system (CNS) involvement or metastasis. In subjects suspected of having CNS disease, a magnetic resonance imaging (MRI) scan of the brain and lumbar puncture should be done to confirm.
* Documented human immunodeficiency virus (HIV), active bacterial infections, active or chronic hepatitis B, hepatitis C.

  * Positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antigen (HBsAb) positive and hepatitis B core antibody (HBcAb) negative) or a fully resolved acute hepatitis B infection is not an exclusion criterion.
  * If hepatitis C antibody test is positive, then the patient must be tested for the presence of hepatitis C virus (HCV) by reverse transcription polymerase chain reaction (RT-PCR) and be HCV ribonucleic acid (RNA) negative

NOTE: HIV-positive patients are excluded from the study. Alemtuzumab may produce a different pattern of toxicities in patients with HIV infection; in addition, the depletion of T cells produced by alemtuzumab may have adverse effects on HIV-positive individuals.

* Concurrent anticancer therapy (including other investigational agents).
* History of severe asthma or presently on chronic inhaled corticosteroid medications (patients with a history of mild asthma not requiring corticosteroid therapy are eligible).
* Patients with smoldering and lymphomatous ATL.
* Pregnant or nursing patients.
* Patients who have previously received alemtuzumab are ineligible. NOTE: Patients with relapsed T-cell prolymphocytic leukemia (T-PLL) who have achieved at least a partial response to prior alemtuzumab are eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, moderate/severe graft versus host disease, cognitive impairment, active substance abuse, or psychiatric illness/social situations that, in the view of the Investigator, would preclude safe treatment or the ability to give informed consent and limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Miljkovic MD, Dubois SP, Muller JR, Bryant B, Ma E, Conlon KC, Waldmann TA. Interleukin-15 augments NK cell-mediated ADCC of alemtuzumab in patients with CD52+ T-cell malignancies. Blood Adv. 2023 Feb 14;7(3):384-394. doi: 10.1182/bloodadvances.2021006440. PMID 35475910
- [Derived] Dubois SP, Miljkovic MD, Fleisher TA, Pittaluga S, Hsu-Albert J, Bryant BR, Petrus MN, Perera LP, Muller JR, Shih JH, Waldmann TA, Conlon KC. Short-course IL-15 given as a continuous infusion led to a massive expansion of effective NK cells: implications for combination therapy with antitumor antibodies. J Immunother Cancer. 2021 Apr;9(4):e002193. doi: 10.1136/jitc-2020-002193. PMID 33883258
- [Derived] Waldmann TA, Dubois S, Miljkovic MD, Conlon KC. IL-15 in the Combination Immunotherapy of Cancer. Front Immunol. 2020 May 19;11:868. doi: 10.3389/fimmu.2020.00868. eCollection 2020. PMID 32508818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0062.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled on Level 3 - 3 mcg/kg/dose of Interleukin 15 (IL-15) Followed by Alemtuzumab.
Groups:
- Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15): IL-15 for 10 doses over two weeks
  IL-15 plus: Recombinant Human IL-15 (subcutaneous (s.c.) rhIL-15) by s.c. injection Monday-Friday over two weeks.
- Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab; Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab: IL-15 for 10 doses over two weeks followed by alemtuzumab for 4 weeks
  IL-15 plus: Recombinant Human IL-15 (subcutaneous (s.c.) rhIL-15) by s.c. injection Monday-Friday over two weeks.
  alemtuzumab: Alemtuzumab three times a week for a total of 4 weeks of alemtuzumab treatment.
Period: Overall Study
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Started | 3 | 4 | 4
Completed | 3 | 3 | 3
Not Completed | 0 | 1 | 1
Not completed — Progressive disease | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Total
Number analyzed (Participants) | 3 | 4 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 9
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.47 (10.71) | 57.1 (14.54) | 47.68 (3.33) | 45.05 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 0 | 1 | 1 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Subcutaneous Recombinant Human IL-15 (s.c. rhIL-15)
Description: MTD is defined as the dose level at which no more than 1 of up to 6 participants experience a dose-limiting toxicity (DLT) during the first 6 weeks of treatment, and the dose below that at which at least 2 (of≤6) participants have DLT as a result of the drug. A DLT is defined as any grade 3 or 4 toxicity possibly, probably or definitely related to the rhIL-15 treatment that occurs during the first 6 weeks of treatment with some exceptions such as grade 3 or 4 lymphopenia, and grade 3 neutropenia for example.
Time Frame: 6 weeks
Measure: Number; unit: mcg/kg/dose
Groups:
- All Participants: All participants who received at least one dose of subcutaneous Recombinant Human IL-15 (s.c. rhIL-15) followed by Alemtuzumab
Arm/Group | All Participants
Number analyzed (Participants) | 11
mcg/kg/dose | 2

2. Primary Outcome: Number of Dose-limiting Toxicities (DLTs) of Subcutaneous Recombinant Human IL-15 (s.c. rhIL-15) Administered With 3 Times Per Week Intravenous (IV) Alemtuzumab
Description: A DLT is defined as any grade 3 or 4 toxicity possibly, probably or definitely related to the rhIL-15 treatment that occurs during the first 6 weeks of treatment with some exceptions such as grade 3 or 4 lymphopenia, and grade 3 neutropenia for example.
Time Frame: 6 weeks
Measure: Number; unit: toxicities
Groups:
- Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab: IL-15 for 10 doses over two weeks followed by alemtuzumab for 4 weeks per dosing schema to determine the maximum tolerated dose (MTD)
  IL-15 plus: Recombinant Human IL-15 (subcutaneous (s.c.) rhIL-15) by s.c. injection Monday-Friday over two weeks.
  alemtuzumab: Alemtuzumab three times a week for a total of 4 weeks of alemtuzumab treatment.
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 3 | 4 | 4
toxicities
  Possibly related | 1 | 0 | 0
  Probably related | 0 | 0 | 0
  Definitely related | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events Possibly, Probably, and/or Definitely Related to Subcutaneous (s.c. rhIL-15) by Grade Who Have Refractory or Relapsed Chronic and Acute Adult T-cell Leukemia (ATL)Cancer
Description: Here is the number of participants with serious adverse events possibly, probably, and/or definitely related to IL-15 (s.c. rhIL-15) by Grade assessed by the Common Terminology Criteria for Adverse Events (CTCAE 5.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 16 months and 14 days for level 1, 18 months and 12 days for level 2, and 14 months and 24 days for level 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 3 | 4 | 4
Participants
  Grade 3 | 1 | 1 | 1
  Grade 4 | 0 | 0 | 1
  Grade 5 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With a Clinical Response
Description: Clinical response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and reported along with a 95% confidence interval. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: At 3 weeks of treatment and again at 6 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 3 | 4 | 4
Participants
  Complete Response | 1 | 0 | 1
  Partial Response | 0 | 1 | 1
  Stable Disease | 1 | 1 | 1
  Progressive Disease | 1 | 2 | 1

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured from the date of protocol consent until death or progressive disease occurs. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and reported along with a 95% confidence interval. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions.
Time Frame: Restaging by computerized tomography (CT) occurred at the end of week 3 and week 6 during treatment, then every 60 days for 6 months, and every 90 days for up to 2 years after finishing treatment.
Measure: Median (Full Range); unit: Days
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 3 | 4 | 4
Days | 78 [42 to 84] | 83 [29 to 412] | 138 [2 to 760]

6. Secondary Outcome: Percentages of Circulating Lymphocytes (T and NK Cells) and the T-cell Subsets
Description: Biological effects of rhIL-15 administered with alemtuzumab on the percentages of circulating lymphocytes (T and NK cells) and the T-cell subsets naïve, central and effector memory subsets (based on expression of cluster of differentiation 52 (CD52), neural cell adhesion molecule (CD56), cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), memory T cells (CD45RO), memory T cells (CD45RA), cluster of differentiation 28 (CD28), apoptosis antigen 1 (CD95), C-C Chemokine Receptor 4 (CD194), C-C Motif Chemokine Receptor 7 (CCR7) and L-selectin (CD62L) using flow cytometry.
Time Frame: At 6 weeks of treatment
Population: These analyses were not performed because there was pan lymphocyte depletion with the initiation of Campath (alemtuzumab) treatment and flow cytometry was not performed and there were not enough circulating lymphocytes to analyze.
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Plasma Levels of Pro-inflammatory Cytokines
Description: Plasma levels of pro-inflammatory cytokines using flow cytometry.
Time Frame: At 6 weeks of treatment
Population: as for outcome 6
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Regardless of Attribution Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events regardless of attribution assessed by the Common Terminology Criteria for Adverse Events (CTCAE 5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
Number analyzed (Participants) | 3 | 4 | 4
Participants | 3 | 4 | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 16 months and 14 days for level 1, 18 months and 12 days for level 2, and 14 months and 24 days for level 3.
Arm/Group | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab (N=3) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab (N=4) | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab (N=4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 - 0.5 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab (N=3) | Level 2 - 1 mcg/kg/Dose of Interleukin-15 (IL-15) Followed by Alemtuzumab (N=4) | Level 3 - 2 mcg/kg/Dose of Interleukin 15 (IL-15) Followed by Alemtuzumab (N=4)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (9) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (4) | 2 (3)
Fever (General disorders) | 2 (3) | 3 (8) | 2 (4)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (5) | 2 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (8) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 1 (1)
Infections and infestations - Other, CMVpositive (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 1 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, CMV positive (Investigations) | 1 (3) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (5) | 3 (7) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, tumor bleeding in left ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (4) | 2 (4) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 2 (9) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02689453/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02689453/ICF_001.pdf